CLINICAL TRIAL: NCT01939522
Title: An Open Label Single-arm Trial of the Immunogenicity and Reactogenicity of a 13-valent Pneumococcal Conjugate Vaccine (Prevenar13®) Given to Children With Type 1 Diabetes Mellitus Who Have Not Previously Received a Primary Schedule of Immunisation With Pneumococcal Conjugate Vaccines in Infancy.
Brief Title: Protection Against Pneumococcal Infection in Children With T1DM
Acronym: T1DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OVG 2013/03; 2013-001024-19 (EudraCT Number)
Record Dates: First submitted 2013-06-04; First posted 2013-09-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; pneumococcal
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevenar13® (13-valent pneumococcal conjugate vaccine) (Experimental): Prevenar13 administered as a single dose, 0.5ml Intramuscular liquid form intervention at baseline.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (PCV13)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (PCV13)
  Other Names: Prevenar13®

SUMMARY:
Children/ young people with diabetes may be at a higher risk of acquiring certain infections. These infections include those caused by a bacterium called the pneumococcus which can cause pneumonia, meningitis and ear infections. In the UK older children with diabetes are given a vaccine against the pneumococcus bug called Pneumovax (or PPS23 for short). Although PPS23 causes a good immune response in children over 2 years of age it is not actually known how well PPS23 protects against infection in children of any age. In addition there is some data in adults and children that PPS23 may result in a reduced response to future doses of pneumococcal vaccines (hyporesponsiveness). Because of the lack of information on how well PPS23 protects and potential hyporesponsiveness the investigators would like to study the use of an alternative vaccine against pneumococcus called Prevenar13 (or pCV13). This vaccine is known to be safe and to work well in babies and young children and there have been no concerns about hyporesponsiveness. It has been approved for use in children up to 17 years of age but there is little information on the size and duration of immune response to PCV13 in children aged 6 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1DM and being followed in the Oxfordshire Children's Diabetes Service.
* Aged between 6 years and 17 years.
* Parent/legal guardian willing and able to give informed consent.
* No previous immunisation with a pneumococcal conjugate vaccine (PCV).
* Willing to allow the General Practitioner to be notified of participation in the study.

Exclusion Criteria:

* Known allergic reaction to the vaccine antigen or any of the excipients.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pneumococcal serotype-specific (SpVS) antibody concentrations at 3 months following a single dose of 13-valent pneumococcal conjugate vaccine (PCV13) | 3 months after vaccination
  The geometric mean concentration (GMC), together with 95% confidence intervals, of SpVS antibody at baseline, 3 months and 12 months following a single dose of PCV13.

SECONDARY OUTCOMES:
Pneumococcal serotype-specific GMC for serotypes 4, 7F & 19A at 3 months after immunisation with a single dose of PCV13 in the children who have had a prior dose of PPS23 vs those who have not. | 3 months after vaccination
  The difference between the pneumococcal serotype-specific geometric mean antibody concentrations (GMC) for serotypes 4, 7F and 19A at three months after immunisation with a single dose of 13-valent pneumococcal conjugate vaccine (PCV13) in the children who have had a prior dose of 23-valent pneumococcal polysaccharide vaccine (PPS23) versus those who have not.
Pneumococcal serotype-specific (SpVS) antibody concentrations at baseline and 12 months following a single dose of 13-valent pneumococcal conjugate vaccine (PCV13). | 12 months after vaccination
  The proportion of children with vaccine pneumococcal serotype-specific (SpVS) antibody concentrations >0.35mcg/ml at baseline and 12 months following a single dose of 13-valent pneumococcal conjugate vaccine (PCV13).
GMC of SpVS antibody at baseline, 3mnth and 12mnth following 1 dose of PCV13 | 12 months after vaccination
  To determine the GMC, together with 95% confidence intervals, of SpVS antibody at baseline, 3mnth and 12mnth following 1 dose of PCV13
Pneumococcal serotype-specific GMC for all vaccine-specific serotypes (VS) at baseline, 3 months and 12 months following immunisation with a single dose of PCV13 in children who have had a prior dose of PPS23 and those who have not. | 12 months after vaccination
  The difference between the pneumococcal serotype-specific GMC for all vaccine-specific serotypes (VS) at baseline, 3 months and 12 months following immunisation with a single dose of PCV13 in children who have had a prior dose of 23-valent pneumococcal polysaccharide vaccine (PPS23) versus those who have not.
Pneumococcal serotype-specific antibody concentrations for all VS in children who have had a prior dose of 23-valent pneumococcal polysaccharide vaccine (PPS23) and those who have not. | 12 months after vaccination
  The difference between the proportion of children with pneumococcal serotype-specific antibody concentrations >0.35mcg/ml for all VS in children who have had a prior dose of 23-valent pneumococcal polysaccharide vaccine (PPS23) versus those who have not.
Vaccine-specific serotype antibody concentration between baseline and 3 months with HbA1C. | 3 months after vaccination
  The correlation coefficient for the increase in VS antibody concentration between baseline and 3 months and HbA1C at baseline.
Blood glucose control in the week preceding and the week following immunisation with PCV13 | One week after vaccination
  A descriptive analysis of blood glucose control in the week preceding and the week following immunisation with PCV13

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom